CLINICAL TRIAL: NCT06896279
Title: Study on the Effectiveness and Safety of Temporal Interference Stimulation in Treating Patients With Severe Consciousness Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai First Rehabilitation Hospital (Unknown)
Responsible Party: Principal Investigator, Xuehai Wu, Deputy Director of Shanghai Neurosurgical Emergency Center, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HY-TI2024-01
Record Dates: First submitted 2025-03-03; First posted 2025-03-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-03

CONDITIONS: Disorder of Consciousness; Temporal Interference Stimulation
Keywords: Disorder of Consciousness; Randomized clinical trail; Temporal Interference Stimulation
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is being conducted as a double-blind trial, wherein the surgeons, assessors and participants' family members are kept unaware of the assigned research groups. However, it is necessary to inform the physicians responsible for adjustment of stimulation parameters about the allocation of participants. Follow-up assessments of participants after stimulation will be conducted by an independent assessor using standardized evaluation criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TI stimulation group (Experimental): The two high-frequency electric fields of the TI device are set at different frequencies, thereby resulting in the generation of a low-frequency electric field that is capable of triggering brain physiological responses. The duration is 10 minutes.
  Interventions: Procedure: TI Stimulation
- Sham TI stimulation group (Sham Comparator): The two high-frequency electric fields of the TI device are set to be completely of the same frequency (2000Hz), thus no low-frequency electric field is produced and no cerebral physiological responses are elicited. The duration lasts for 10 minutes.
  Interventions: Procedure: Sham Stimulation

INTERVENTIONS:
Procedure: TI Stimulation — Participants will accept the TI stimulus for one month
  Arms: TI stimulation group
Procedure: Sham Stimulation — Participants will accept the sham TI stimulus for one month
  Arms: Sham TI stimulation group

SUMMARY:
Investigating the efficacy and safety of temporal interference stimulation for patients with disorders of consciousness.

DETAILED DESCRIPTION:
Based on the central loop hypothesis, deep brain stimulation (DBS) represents a commonly utilized neuro-modulation stimulation technology for disorders of consciousness (DOC). It was initially employed in Europe in 1968 for treating DOC. Some patients can regain functional communication capabilities and even resume family life. Nevertheless, as a neurosurgical intervention, DBS implantation entails significant surgical risks and potential complications (such as cerebral edema in the surgical area, secondary cerebral hemorrhage, secondary epilepsy, postoperative brain abscess, pulse generator shutdown or circuit malfunction, displacement of stimulation electrodes or extension leads, rejection reactions), and incurs substantial costs, imposing a heavy burden on patients' families and the national medical insurance fund. Traditional non-invasive brain stimulation methods, such as transcranial alternating or direct current stimulation, although not requiring surgery, have limited focusing capacity and the ability to stimulate deep brain structures. Hence, researchers have been in pursuit of approaches to precisely and effectively stimulate deep brain regions without the need for surgery.

In 2017, the concept of temporal interference (TI) stimulation, a novel non-invasive method for regulating deep brain regions was put forward . The fundamental principle of TI stimulation is that two interfering high-frequency signals will generate a low-frequency amplitude-modulated electric field, which can drive the discharge of deep brain neurons. Furthermore, by fixing the sum of the input currents of two pairs of electrodes and altering the current input ratio of the two pairs of electrodes, the movement of the mouse's forepaws, whiskers, and ears without modifying the spatial position of the electrodes could be achieved. Therefore, TI stimulation enables the flexible movement of the stimulation target area within the brain without electrode displacement. Despite the fact that research on TI technology is still in its nascent stage, this method has demonstrated substantial potential in neuroscience and clinical therapy.

Consequently, the objective of this multicenter randomized controlled trial is to assess the therapeutic effect of temporal interference stimulation in awakening patients with severe disorders of consciousness and verify its safety. Simultaneously, it aims to clarify issues such as the clinical application indications, operational parameters of TI. This will facilitate a deeper comprehension of the effectiveness, clinical application indications, operational parameters, and treatment plans of this emerging neuro-modulation technology as a means of awakening treatment, and promote the advancement of diagnosis and treatment technologies for patients with severe disorders of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Severe consciousness disorder patients aged 18 to 75 years old, regardless of gender;
* Patients with severe consciousness disorders, namely a minimally conscious state or vegetative state that lasts for 28 days or more;
* Patients with normal body temperature, stable vital signs, spontaneous breathing, tracheotomy without the use of a metal cannula and with a small amount of sputum, and who are eligible for magnetic resonance imaging (MRI) examination;
* Written informed consent obtained from the patient's family members in advance.

Exclusion Criteria:

* Individuals with a previous history of significant neuropsychiatric and other major disorders such as those involving the heart, lung, liver, and kidney;
* Those who have undergone V-P shunt or Ommaya reservoir implantation and other procedures that may influence the analysis of magnetic resonance scanning signals;
* Patients who are scheduled for V-P shunt or Ommaya reservoir implantation in the near future;
* Pregnant women;
* Those who have participated in other drug or device clinical trials;
* Patients with poorly controlled epilepsy in the recent period;
* Those with infections at the TI stimulation site or compromised skin integrity at the electrode placement site;
* Those currently taking medications prone to inducing epilepsy, such as quinolone drugs;
* Those with intracranial infections, intracranial tumors, or metallic objects within the cranium;
* Those allergic to electrode gel or adhesives;
* Those with implanted electronic devices within the body;
* Those with severe cardiac disorders and those equipped with cardiac pacemakers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Effective rate of awakening | Stimulation for 1 month
  The CRS-R is employed, with a minimum of 5 CRS-R assessments conducted at each follow-up time point, accompanied by simultaneous video recording. And the highest value is scored as a state of consciousness. The clinical assessment of participants' consciousness is deemed significantly improved when it fulfills the following criteria: a) MCS- recover to consciousness level of MCS+ or higher; b) Vegetative state(VS) recover to consciousness level of MCS- or higher; c) MCS status (MCS- or MCS+) recover to emergence from MCS (restoration of functional communication).

SECONDARY OUTCOMES:
The difference of CRS-R scale relative to baseline between TI group and sham group | Stimulation begin for 14 days, 1 month and 3 months
  The Coma Recovery Scale-Revised (CRS-R) is a standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness. It has good validity, reliability and practicability.
The difference of Simplified Evaluation of CONsciousness Disorders (SECONDs) scale relative to baseline between TI group and sham group | Stimulation begin for 14 days, 1 month and 3 months
  The SECONDs is a fast tool to assess consciousness in brain-injured patients. The minimum score is 0 and the maximum is 8, higher scores mean a better outcome.
The difference of modified Ashworth scale relative to baseline between TI group and sham group | Stimulation begin for 14 days, 1 month and 3 months
  The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone. The minimum grade is 0 and the maximum is 4, higher scores mean a worse outcome.
The difference of Nociception Coma Scale-Revised (NCS-R) scale relative to baseline between TI group and sham group | Stimulation begin for 14 days, 1 month and 3 months
  The NCS-R was developed to help assess pain in patients with disorders of consciousness (DOC). Several studies have shown its sensitivity in assessing response to acute noxious stimuli. The minimum score is 0 and the maximum is 12, higher scores mean a better outcome.
The difference of effective rate of awakening between TI group and sham group by CRS-R scale | Stimulation begin for 1 month and 3 months
  The Coma Recovery Scale-Revised (CRS-R) is a standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness. It has good validity, reliability and practicability.
The difference of effective rate of awakening between TI group and sham group by Simplified Evaluation of CONsciousness Disorders (SECONDs) scale | Stimulation begin for 1 month and 3 months
  The SECONDs is a fast tool to assess consciousness in brain-injured patients. The minimum score is 0 and the maximum is 8, higher scores mean a better outcome.
The difference of recovery trajectories of consciousness level between TI group and Sham group | Stimulation for 3-month-stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Xuehai Wu, Ph.D., Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University
Locations (2):
- China (2):
  - Department of neurological rehabilitation, Shanghai First Rehabilitation Hospital, Tongji University, Shanghai, Shanghai Municipality
  - Department of Neurosurgery, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Nov;26(11):1994-2004. doi: 10.1038/s41593-023-01456-8. Epub 2023 Oct 19. Erratum In: Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. PMID 37857775
- [Result] Thibaut A, Schiff N, Giacino J, Laureys S, Gosseries O. Therapeutic interventions in patients with prolonged disorders of consciousness. Lancet Neurol. 2019 Jun;18(6):600-614. doi: 10.1016/S1474-4422(19)30031-6. Epub 2019 Apr 16. PMID 31003899
- [Result] Giacino JT, Katz DI, Schiff ND, Whyte J, Ashman EJ, Ashwal S, Barbano R, Hammond FM, Laureys S, Ling GSF, Nakase-Richardson R, Seel RT, Yablon S, Getchius TSD, Gronseth GS, Armstrong MJ. Practice guideline update recommendations summary: Disorders of consciousness: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; the American Congress of Rehabilitation Medicine; and the National Institute on Disability, Independent Living, and Rehabilitation Research. Neurology. 2018 Sep 4;91(10):450-460. doi: 10.1212/WNL.0000000000005926. Epub 2018 Aug 8. PMID 30089618
- [Result] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- [Result] Tasserie J, Uhrig L, Sitt JD, Manasova D, Dupont M, Dehaene S, Jarraya B. Deep brain stimulation of the thalamus restores signatures of consciousness in a nonhuman primate model. Sci Adv. 2022 Mar 18;8(11):eabl5547. doi: 10.1126/sciadv.abl5547. Epub 2022 Mar 18. PMID 35302854
- [Result] Schiff ND. Recovery of consciousness after brain injury: a mesocircuit hypothesis. Trends Neurosci. 2010 Jan;33(1):1-9. doi: 10.1016/j.tins.2009.11.002. Epub 2009 Dec 1. PMID 19954851